CLINICAL TRIAL: NCT03613428
Title: Phase I/II Study of Ruxolitinib Plus L-asparaginase, Vincristine, and Prednisone in Adult Patients With Relapsed or Refractory Early T Precursor Acute Lymphocytic Leukemia
Brief Title: Ruxolitinib Plus LVP in Patients With R/R ETP-ALL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Clinical Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-ETP-01
Record Dates: First submitted 2018-07-16; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Acute T Cell Leukemia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — ruxolitinib; Vincristine; Prednisone; Steroids

STUDY DESIGN:
Intervention Model Description: Open label dosing cohorts will evaluate oral ruxolinitib (doses ranging from 10 - 80 mg) in combination with vincristine (1.4 mg/m2) and oral prednisone (1 mg/kg, 5 days a week for 4 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ruxolitinib, vincristine, prednisone (Experimental): Open label dosing cohorts will evaluate oral ruxolitinib (doses ranging from 10 - 80 mg) in combination with vincristine (1.4 mg/m2) and oral prednisone (1 mg/kg, 5 days a week for 4 weeks).
  Interventions: Drug: Ruxolitinib; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Ruxolitinib — Dose escalation up to 80 mg administered orally
  Other Names: JAK1/JAK2 inhibitor
Drug: Vincristine — 1.4 mg/m2 i.v. weekly for 4 weeks
  Other Names: Oncovin
Drug: Prednisone — 1 mg/kg orally 5 consecutive days per week for 4 weeks.
  Other Names: steroid

SUMMARY:
To determine the maximum tolerated dose (MTD), if present, and dose schedule of ruxolitinib in combination with L-ASP, vincristine, and prednisone (LVP) in patients with relapsed-and-refractory (R/R) early T precursor acute lymphocytic leukemia (ETP-ALL). Once determined, the purpose of this study will be to determine the efficacy of ruxolitinib in combination with LVP in patients with R/R ETP-ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with early T-precursor ALL, with any of the following:

   * refractory to primary induction therapy or refractory to salvage therapy,
   * in untreated first relapse with first remission duration <12 months
   * in untreated second or greater relapse
   * relapse at any time after allogeneic HSCT
2. Subject has received intensive combination chemotherapy for the treatment of ALL for initial treatment or subsequent salvage therapy.
3. Greater than 5% blasts in the bone marrow
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

1. Malignancy other than ALL within 5 years before recruitment, except for adequately treated selected cancers without evidence of disease
2. Current relevant central nervous system (CNS) pathology or known or suspected CNS involvement
3. Isolated extramedullary disease
4. Current autoimmune disease or history of autoimmune disease with potential CNS involvement
5. Autologous HSCT within 6 weeks or allogeneic HSCT within 12 weeks before blinatumomab treatment, or eligibility for allogeneic HSCT at the time of enrollment
6. Active acute grade 2 to 4 graft versus host disease (GvHD) according to Glucksberg et al (1974) criteria that required systemic treatment to prevent or treat GvHD 2 weeks before blinatumomab treatment
7. Known exclusion criteria to investigator choice of SOC chemotherapy (per package insert)
8. Cancer chemotherapy or radiotherapy with 2 weeks, or immunotherapy (included CD19 therapy) within 4 weeks of protocol-specified therapy
9. Abnormal laboratory values (alanine or aspartate transaminase [ALT or AST] or alkaline phosphatase [ALP] ≥ 5 × upper limit of normal [ULN]; total bilirubin or creatinine ≥ 1.5 × ULN), or calculated creatinine clearance < 60 mL/min.

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Establish optimal dose of ruxolitinib | Upon completion of a 28 day treatment cycle
  Determine maximum tolerated dose (MTD) of ruxolitinib

SECONDARY OUTCOMES:
Evaluate safety by assessing toxicities | Upon completion of a 28 day treatment cycle
  Evaluate safety by assessing possible toxicities of thrombocytopenia, neutropenia, serum creatinine, total bilirubin, diarrhea, and/or vomiting.
Overall response | At the end of Cycle 2 (each cycle is 60 days)
Complete response | At the end of Cycle 2 (each cycle is 60 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ji, MD, Principal Investigator — West Chinia Hospital, Sichuan University